CLINICAL TRIAL: NCT01078051
Title: Drug-Eluting Stent Implantation Versus Optimal Medical Treatment in Patients
Brief Title: Drug-Eluting Stent Implantation Versus Optimal Medical Treatment in Patients With Chronic Total Occlusion (DECISION-CTO)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: at sponsor's discretion : Benefit is not guaranteed
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0647
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
Keywords: chronic total occlusion; stent; medical therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimal medical therapy (Active Comparator): optimal medical therapy
  Interventions: Drug: optimal medical therapy
- drug-eluting stent (Active Comparator): Cypher, xience, Endeavor, Taxus
  Interventions: Procedure: Cypher, xience, Endeavor, Taxus

INTERVENTIONS:
Procedure: Cypher, xience, Endeavor, Taxus — all species of drug-eluting stent implantation
  Other Names: percutaneous coronary intervention
  Arms: drug-eluting stent
Drug: optimal medical therapy — optimal medical therapy
  Other Names: intensive medical therapy
  Arms: Optimal medical therapy

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of drug-eluting stent implantation compared to optimal medical treatment in patients with chronic total occlusion.

DETAILED DESCRIPTION:
Prospective, two arms, randomized multi-center trial in Asian-pacific region. Following angiography, patients with chronic total occlusion (more than 3 months) have documented myocardial ischemia or symptoms of angina, and eligible for stenting without any exclusion criteria will be randomized 1:1 to: a) drug-eluting stent vs. b) optimal medical treatment. All patients will be followed for at least 3 year.

The subjects with chronic total occlusion but failed to random for any reason, they will be enrolled in registry group.

The random design was closed at the date of 22 July 2019 however already randomized subjects and subjects from registry design continue 10 years follow-up on IRIS-CTO registry.

ELIGIBILITY:
Inclusion Criteria:

Clinical

1. Patients with angina or silent ischemia and documented ischemia
2. Patients who are eligible for intracoronary stenting
3. Age > 18 years

Angiographic

1. De novo lesion CTO
2. Reference vessel size 2.5 mm by visual estimation
3. At least one CTO lesions located in proximal or mid epicardial coronary artery. (If the patient has two CTO lesions, one CTO lesion should be located in proximal or mid epicardial coronary artery)

CTO definition: TIMI flow 0 and estimated duration over 3 months The duration of the occlusion was determined by the interval from the last episode of acute coronary syndrome, or In patients without a history of acute coronary syndrome, from the first episode of effort angina consistent with the location of the occlusion

1. Angiographically defined total occlusion over 3 months
2. If no definite symptom with total occlusion, two experienced operators decide CTO in consideration of angiographical morphology (degree of calcification, bridging collaterals, non-tapered stump, angiographic filling from collaterals)

Exclusion Criteria:

1. History of bleeding diathesis or coagulopathy
2. Pregnant state
3. Three vessel CTO
4. Known hypersensitivity or contra-indication to contrast agent and heparin
5. ST-elevation acute myocardial infarction requiring primary stenting
6. Characteristics of lesion 1) Left main disease 2) In-stent restenosis 3) Graft vessels 4) Distal epicardial coronary artery CTO lesions
7. Hematological disease
8. Hepatic dysfunction, liver enzyme (ALT and AST) elevation 3 times normal
9. Renal dysfunction, creatinine more than 2.0
10. Contraindication to aspirin, clopidogrel or other commercial antiplatelet agent
11. Left ventricular ejection fraction
12. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
13. Non-cardiac co-morbid conditions are present with limited life expectancy or that may result in protocol non-compliance (per site investigator's medical judgment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 2010-03-22 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Composite outcomes of all cause death, myocardial infarction, stroke, and any revascularization for 3 years after randomization | at 3 years
  at the median of 3 years

SECONDARY OUTCOMES:
All Death (Cardiac death) | at 3 years & 5 years
Angina class; Quality of life, clinical outcomes at 5 years | at 3 years & 5 years
Myocardial infarction, stroke,any revascularization, CTO-vessel related revascularization, hospitalization due to acute coronary syndrome, left ventricular ejection fraction | at 3 years & 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD,PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (26):
- Ruby Hall Clinic, Pune, India
- Medistra Hospital, Jakarta, Indonesia
- South Korea (21):
  - Sam Anyang Hospital, Anyang
  - Soonchunhyang University Hospital, Buchen, Bucheon-si
  - Soonchunhyang University Hospital, Cheonan, Cheonan
  - Chungbuk National University Hospital, Cheongju-si
  - Kangwon National University Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon ST.Mary's Hospital, Daejeon
  - GangNeung Asan Hospital, Gangneung
  - Chonbuk National University Hospital, Jeonju
  - Chonnam National University Hospital, Kwangju
  - Dong-A University Medical Center, Pusan
  - Pusan National University Yangsan Hospital, Pusan
  - Asan Medical Center, Seoul
  - Hallym University Medical Center, Hangang Sacred Heart Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea, Kangnam ST.Mary's Hospital, Seoul
  - Bundang CHA Hospital, Sŏngnam
  - Ulsan University Hospital, Ulsan
  - Wonju Christian Hospital, Wŏnju
- Taiwan (2):
  - National Taiwan University hospital, Taipei
  - Shin Kong Hospital, Taipei
- King chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.

REFERENCES:
- [Derived] Lee SW, Lee PH, Ahn JM, Park DW, Yun SC, Han S, Kang H, Kang SJ, Kim YH, Lee CW, Park SW, Hur SH, Rha SW, Her SH, Choi SW, Lee BK, Lee NH, Lee JY, Cheong SS, Kim MH, Ahn YK, Lim SW, Lee SG, Hiremath S, Santoso T, Udayachalerm W, Cheng JJ, Cohen DJ, Muramatsu T, Tsuchikane E, Asakura Y, Park SJ. Randomized Trial Evaluating Percutaneous Coronary Intervention for the Treatment of Chronic Total Occlusion. Circulation. 2019 Apr 2;139(14):1674-1683. doi: 10.1161/CIRCULATIONAHA.118.031313. PMID 30813758
- [Derived] Azzalini L, Vo M, Dens J, Agostoni P. Myths to Debunk to Improve Management, Referral, and Outcomes in Patients With Chronic Total Occlusion of an Epicardial Coronary Artery. Am J Cardiol. 2015 Dec 1;116(11):1774-80. doi: 10.1016/j.amjcard.2015.08.050. Epub 2015 Sep 11. PMID 26434510